CLINICAL TRIAL: NCT05493306
Title: Evaluation Der Telerehabilitation im Anschluss an Eine stationäre Oder Ambulante Rehabilitation Phase II - Pilotprojekt [Evaluation of Telerehabilitation Following Inpatient or Outpatient Rehabilitation Phase II - Pilot Project]
Brief Title: Evaluation of Telerehabilitation Following Inpatient or Outpatient Rehabilitation Phase II
Status: Completed | Type: Observational
Sponsor: Pensionsversicherungsanstalt (Other)
Responsible Party: Sponsor
Other Study IDs: 0002 Evaluation Telereha
Record Dates: First submitted 2022-08-05; First posted 2022-08-09 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-07

CONDITIONS: Oncology; Musculoskeletal Diseases
Keywords: Telerehabilitation; Evaluation; Usability
MeSH Terms: conditions — Neoplasms; Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Telerehabilitation is implemented in the Pensionsversicherungsanstalt (PVA) as an independent rehabilitation offer following a rehabilitation phase II. This offer primarily includes physiotherapeutic training units in group settings and in individual counselling, as well as health-related educational sessions and doctor's consultations via video conferencing, initially for rehabilitation patients with diseases of the musculoskeletal system or oncological diseases. The first stage of the implementation process was evaluated with a focus on acceptance, usability and feasibility from the perspective of patients and treatment team.

The evaluation was based on a convergent mixed methods design (Creswell & Plano Clark, 2017) to draw on the strengths of qualitative and quantitative research approaches (Creswell & Creswell, 2018). Qualitative and quantitative data were generated in parallel and treated equally. The perspective of the patients (N = 86) was collected through online questionnaires and in-depth telephone interviews (N = 22) and that of the treatment team through a questionnaire survey (N = 32) and focus group interviews (N = 24). The administrative team (N = 8) was asked for their assessment in a focus group interview. Technical difficulties in the implementation of telerehabilitation were documented by the treatment team. The consolidation of these multi-perspective results took place at the level of interpretation.

ELIGIBILITY:
Inclusion Criteria:

Patients who have completed rehabilitation (phase II) with the indications:

* musculoskeletal diseases
* oncology.

Exclusion Criteria:

* Failure to obtain the declaration of consent
* Lack of the required technical aids (mobile phone, tablet or PC)
* Lack of the technical skills to operate the app and thus to participate in telerehabilitation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have completed rehabilitation phase II and have been assessed by their doctor as suitable for telerehabilitation. Involved treatment team and administrative team.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Usability of the telerehabilitation | April 2021 - May 2022
  The patients' perspective was collected with a self-developed online questionnaire (N = 86) and in-depth telephone interviews (N = 22).
  The questionnaires were analysed descriptively. The telephone interviews were protocolled and subsequently coded and categorised.
  The perspective of the treatment team was collected with a self-developed questionnaire (N = 32) and focus group interviews (N = 24).
  In addition, the administrative team (N = 8) was asked for their assessments in a focus group interview. The questionnaires were analysed descriptively. The focus group interview was recorded and subsequently coded and categorised.
Feasibility of the telerehabilitation | April 2021 - May 2022
  Technical difficulties concerning the video calls were continuously documented by the treatment team. The data were analysed descriptively.
Acceptance of the telerehabilitation | April 2021 - May 2022
  The patients' perspective was collected with a self-developed online questionnaire (N = 86) and in-depth telephone interviews (N = 22).
  The questionnaires were analysed descriptively. The telephone interviews were protocolled and subsequently coded and categorised.
  The perspective of the treatment team was collected with a self-developed questionnaire (N = 32) and focus group interviews (N = 24).
  The questionnaires were analysed descriptively. The focus group interviews were recorded and subsequently coded and categorised.

CONTACTS AND LOCATIONS:
Overall Officials: David Felder, Mag., Study Chair — Pensionsversicherungsanstalt
Locations (1):
- PVA - Zentrum für ambulante Rehabilitation Graz, Graz, Styria, Austria